CLINICAL TRIAL: NCT02688972
Title: The Accumulative Effect of Cold Water Immersion in Football Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Scheila Marisa Pinheiro (Other)
Responsible Party: Sponsor-Investigator, Scheila Marisa Pinheiro, Student of Master degree, Universidade Federal do Rio Grande do Norte
Organization: Universidade Federal do Rio Grande do Norte (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 861.084
Record Dates: First submitted 2016-02-18; First posted 2016-02-23 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Athletic Performance
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cold water immersion (Experimental)
  Interventions: Other: cold water immersion
- control (Other): 13 volunteers
  Interventions: Other: Control group

INTERVENTIONS:
Other: cold water immersion — The volunteers stayed immerged up to the iliac crest, in the water with water. The temperature utilized was 10 degree C and the time was 10 minutes
  Arms: cold water immersion
Other: Control group — The volunteers stayed in rest about 10 minutes
  Arms: control

SUMMARY:
Football is a sport with congested calendars, which requires muscle recovery strategies such as cold water immersion (CWI). This recovery technique is well spread through football clubs, although it lacks a profound physiologic investigation to understand its effects on athlete's body. Objectives: The main objective of this study is to evaluate the effect of a long-term CWI exposure in football athlete's.

Study Hypothesis:

H0: The application of Cold water immersion doesn't amend the biomarkers, electromyograph signal, power and perceived of recover when compared with control sample.

H1: The application of Cold water immersion amends the biomarkers, electromyograph signal, power and perceived of recover when compared with control sample.

DETAILED DESCRIPTION:
In order to answer this question, the investigators performed a randomized clinical trial in 23 sub-20 football athletes. All subjects were randomly divided into two groups; a control group (10 minutes seated rest) and a CWI group (10 minutes in a 10 degree C) during seven days in a row. The investigators evaluated creatine kinase (CK) and lactate dehydrogenase (LDH) as molecular biomarkers for muscle damage. The blood samples were collected on the first, second, ninth and tenth days. Yet, the investigators assessed the peak of muscle activity and isometric strength of the knee flexors and extensors, potency of lower limbs, perceived exertion (PE) and total quality recovery perceived (TQRPer) in order to understand the treatment physiological effect on the subjects on the first and last day of experiments (before and after training).

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* Soccer players

Exclusion Criteria:

* Neurological, vascular or systemic muscle disease

Ages: 17 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 27 (Actual)
Dates: Start 2015-07; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Biochemical Markers: Creatine Kinase | 10 days
  The creatine kinase was evaluated though blood samples.